CLINICAL TRIAL: NCT02686255
Title: Hemoglobin Trend in Neonates and Toddlers Post Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0655-15-RMC
Record Dates: First submitted 2016-01-28; First posted 2016-02-19 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Congenital Cardiac Defects
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Blood Cell Count

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children 0-18 months post heart surgery: complete blood count for all children 0-18 months going through cardiac surgery
  Interventions: Other: complete blood count

INTERVENTIONS:
Other: complete blood count — complete blood count during follow up in the heart institute

SUMMARY:
Many toddlers and children are released home with relatively low hemoglobin levels following cardiac surgery, and with no careful follow up, at an age at which anemia is common. At this age, breast milk and its substitute do not provide enough iron, and parents are not adherent enough to iron supplements. Due to these facts, there is high importance, especially in children suffering from heart defects, for close follow up on their hemoglobin levels. Studies following hemoglobin trend post cardiac surgery were never done with children.

DETAILED DESCRIPTION:
For the past 6 decades, children have been going through cardiac surgery to correct congenital heart defects. Over the years, there has been great improvement in morbidity and mortality post cardiac surgery due to better technical skill and post operative treatment. Most of those surgeries require cardio-pulmonary bypass machine, which requires the use of blood products, and many of those children also require blood product as part of the post operative care, especially those children with cyanotic heart defects. Many toddlers and children are released home with relatively low hemoglobin levels, and with no careful follow up, at an age at which anemia is a risk factor for developmental delay and decreased cognitive function. Iron deficiency is common in Israel among children aged 6-24 months. At this age, breast milk and its substitute do not provide enough iron, and parents are not adherent enough to iron supplements as recommended by the ministry of health. Due to these facts, there is high importance, especially in children suffering from heart defects, for close follow up on their hemoglobin levels. In adults, a study following hemoglobin levels post cardiac surgery during hospitalization only, showed that most (79%) starting showing improvement during their hospitalization. Another study in patients over the age of 50 post coronary artery bypass graft, showed no difference between a group receiving iron supplements and another not receiving any, after 2 months. Similar studies were never done with children.

ELIGIBILITY:
Inclusion Criteria:

* All children 0-18 months going through cardiac surgery during the 3 years of the study, after obtaining written consent from the parents/legal guardians.

Exclusion Criteria:

* None

Max Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children 0-18 months going through cardiac surgery during the 3 years of the study
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Hemoglobin levels (mg/dL) during follow up of cardiac surgery, sampled by finger prick | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Gilad Sherman, MD, Principal Investigator — Schneider's children medical center of Israel
Locations (1):
- Rabin medical center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No